CLINICAL TRIAL: NCT06243744
Title: Histological Evaluation of Human Skin Biopsies to Assess the Effects of Renuvion APR Treatment as an Adjunct Procedure in Facelift Surgery
Brief Title: Histological Evaluation of Human Skin Bx to Assess the Effects of APR Tx as an Adjunct Procedure in Facelift Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-21-04
Record Dates: First submitted 2023-12-18; First posted 2024-02-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Skin Laxity; Tissue Degeneration; Tissue Breakdown; Collagen Degeneration; Collagen Shrinkage
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm, study of up to 10 study subjects undergoing a lower facelift surgery and treatment with the Renuvion APR System. The study will be conducted at up to three (3) investigational centers in the United States.
  Two biopsy tissue samples will be taken during the facelift procedure prior to use of the Renuvion APR System and then at the Day 180 visit. Tissue samples will be assessed via microscopy, histology, and immunohistochemistry for biological markers of elasticity (collagen density, elastin, fibrillin-1) and hydration ([aquaporin-3, acidic glycosaminoglycans (GAGs), HA]). Additionally, DNA methylation will be measured in tissue samples to estimate the biological age of the skin.
  Follow-up will occur 1 day, 2 days (optional), 7 days, 14 days, 45 days, 90 days, and 180 days post-procedure with images and skin quality measurements taken as described.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Procedure with the Renuvion APR System in lower facelift area (Other): Subjects will receive a lower facelift surgery per the Investigator's standard clinical practice and treatment with the Renuvion APR System.
  Interventions: Device: Renuvion APR System

INTERVENTIONS:
Device: Renuvion APR System — The Apyx Medical Corporation Renuvion/J-Plasma helium plasma family of products has received FDA clearance under 510(k) numbers K191542, K192867 for the cutting, coagulation, and ablation of soft tissue.

SUMMARY:
The goal of this prospective, single-arm clinical study is to gather quantifiable data on Renuvion's impact on skin elasticity and hydration, indicators of skin quality and estimate the biological skin age using DNA methylation in males and females between 18 and 75 years of age who plan to receive a lower facelift surgery. The main purpose is to quantify the effect of the Renuvion device on skin elasticity (collagen density, elastin, fibrillin-1), hydration (aquaporin-3, acidic glycosaminoglycans, HA), and DNA methylation to estimate the biological age of the skin.

Participants will receive a lower facelift surgery per the Investigator's standard clinical practice and treatment with the Renuvion APR System.

DETAILED DESCRIPTION:
The purpose of this study is to gather quantifiable data on Renuvion's impact on skin elasticity and hydration, indicators of skin quality and estimate the biological skin age using DNA methylation.

This study is a prospective, single-arm clinical study to be conducted at up to three clinical sites in the US. Up to 10 subjects will be enrolled and treated if they meet the inclusion/exclusion criteria and provide written informed consent.

Enrolled subjects meeting all entrance criteria and confirmed eligible for study treatment will be asked to participate. Subjects will receive a lower facelift surgery per the Investigator's standard clinical practice and treatment with the Renuvion APR System. The mid/upper-face area will not be treated with Renuvion and the lower face/neck area will be treated with Renuvion. Treatment will consist of subdermal coagulation of soft tissue using the Renuvion APR handpiece.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ages 18 - 75 years old.
* ASA Physical Status Classification System Class I and Class II subjects.
* Planning to undergo a lower facelift procedure, with or without a neck lift, at the investigator's site.
* Understands and accepts the obligation not to undergo any other procedures or treatments in the areas to be treated during study participation.
* Absence of physical conditions unacceptable to the investigator.
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
* Willing and able to comply with protocol requirements, including study-required images/photos, assessments/measurements, and returning for follow-up visits.
* Willing to release rights for the use of study photos, including in publication.
* Able to read, understand, sign, and date the informed consent.
* Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.

Exclusion Criteria:

* Subjects presenting with ASA Physical Status Classification System Classes III or higher.
* Pregnant, lactating, or plans to become pregnant during study participation.
* Known hypersensitivity or allergy to tumescent anesthetic (lidocaine/ epinephrine).
* Known hypersensitivity or allergy to ibuprofen or other NSAIDS.
* Active systemic or local skin disease that may alter wound healing.
* Significant or uncontrolled medical condition that in the opinion of the investigator participation in the study may compromise the patient's health.
* History of autoimmune disease (excluding Hashimoto's thyroiditis).
* Known susceptibility to keloid formation or hypertrophic scarring.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Possesses a surgically implanted electronic device (i.e. pacemaker).
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Participation in any other investigational study within 30 days prior to consent and throughout study participation.
* Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.
* Subject who has had a prior facelift, neck lift, or Renuvion treatment in the face/neck area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Analysis of Elasticity (collagen density, elastin, & fibrillin-1) | Baseline, Day 180
  To assess Elasticity (collagen density, elastin, & fibrillin-1) evaluation will be based on the qualitative microscopic observation of the stained sections comparing baseline samples to follow-up samples. Histology and immunohistochemistry (IHC) part of the study will be assessed semi-quantitatively. Thus, there will not be units of measurement e.g., weight and height for these evaluations.
  Semi-quantitative scoring for any microscopic changes (H&E staining) and enhancing collagen production (e.g., trichrome staining).
  Four-point Severity Scale Semi-Quantitative Grading of Changes in Histology Samples Description - Definition Normal - Tissue is considered to be normal Minimal - The amount of change present barely exceeds normal limits. Mild (Slight) - The amount of change is easily identified but limited severity. Moderate - The amount of change is prominent, but significant potential for increased severity.
  Severe - The degree of change is as complete as possible
Analysis of Hydration (aquaporin-3, acidic glycosaminoglycans (GAGs), hyaluronic acid (HA)) | Baseline, Day 180
  To assess Hydration (aquaporin-3, GAGs, HA), evaluation will be based on the qualitative microscopic observation of the stained sections comparing baseline samples to follow-up samples. Histology and immunohistochemistry (IHC) part of the study will be assessed semi-quantitatively. Thus, there will not be units of measurement e.g., weight and height for these kinds of evaluations.
  Semi-quantitative scoring for any microscopic changes (H&E staining) and enhancing collagen production (e.g., trichrome staining).
  Four-point Severity Scale Semi-Quantitative Grading of Changes in Histology Samples Description - Definition Normal - Tissue is considered to be normal Minimal - The amount of change present barely exceeds normal limits. Mild (Slight) - The amount of change is easily identified but limited severity. Moderate - The amount of change is prominent, but significant potential for increased severity.
  Severe - The degree of change is as complete as possible
Analysis of Adverse Events | Treatment, Day 1, 7, 14, 45, 90, 180
  Analysis of adverse events through the 180-day post-treatment visit.
Analyzing days of duration for Bruising, Swelling | Post-Treatment, Day 1, 7, 14, 45, 90, 180
  Analysis days of duration of bruising and swelling post-treatment through the 180-day visit.
Days to healed percentage | Post-Treatment, Day 1, 7, 14, 45, 90, 180
  Analysis average number of days to healed profile post-procedure through the 180-day post-treatment visit through Case Report Forms through percentage healed at each follow-up.
Bleeding | During Procedure (Day 0)
  Analysis of bleeding during surgery measured in cubic centimeter.
The Principal Investigator will complete a PGAIS assessing overall aesthetic improvement in the treatment area at day 45, 90, and 180 post-treatment. | Day 45, 90 and180
  Global Aesthetic Improvement Scale Evaluation (PGAIS) rating by investigator [Very much improved, Much improved, Improved, No change, Worse, Much Worse, Very much Worse]
The subject will complete a SGAIS assessing overall aesthetic improvement in the treatment area at day 45, 90, and 180 post-treatment. | Day 45, 90 and180
  Subject Global Aesthetic Improvement Scale Evaluation (SGAIS) rating by subject [Very much improved, Much improved, Improved, No change, Worse, Much Worse, Very much Worse]
Patient Satisfaction | Day 180
  The subject will complete a Patient Satisfaction Questionnaire (PSQ) while referring to their image in a mirror and current post-treatment photos compared to baseline photos to rate how satisfied they are, and if they note any improvement in the treatment area.
Estimated biological age by DNA methylation. | Baseline, Day 180
  DNA methylation (DNAm) will be used to measure the tissue samples to estimate the biological age of the skin. A highly accurate skin-specific age algorithm will analyze these modifications related to human skin health and molecular aging - quantifying the skin health/skin age of the tissue beyond the chronological age of the subject. Hallmarks of aging include genomic instability, telomere attrition, epigenetic alterations, loss of proteostasis, deregulated nutrient sensing, mitochondrial dysfunction, cellular senescence, stem cell exhaustion, and altered intercellular communication.

CONTACTS AND LOCATIONS:
Overall Officials: David Holcomb, M.D., Principal Investigator — Holcomb & Kreithen Plastic Surgery and MedSpa; Melinda Lacerna, M.D., Principal Investigator — LA Plastic Surgery & Dermatology
Locations (2):
- United States (2):
  - LA Plastic Surgery and Dermatology, Bradenton, Florida
  - Holcomb & Kreithen Plastic Surgery and MedSpa, Sarasota, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg SN, Gazelle GS, Halpern EF, Rittman WJ, Mueller PR, Rosenthal DI. Radiofrequency tissue ablation: importance of local temperature along the electrode tip exposure in determining lesion shape and size. Acad Radiol. 1996 Mar;3(3):212-8. doi: 10.1016/s1076-6332(96)80443-0. PMID 8796667
- [Background] Thomsen S. Pathologic analysis of photothermal and photomechanical effects of laser-tissue interactions. Photochem Photobiol. 1991 Jun;53(6):825-35. doi: 10.1111/j.1751-1097.1991.tb09897.x. PMID 1886941
- [Background] Ross EV, McKinlay JR, Anderson RR. Why does carbon dioxide resurfacing work? A review. Arch Dermatol. 1999 Apr;135(4):444-54. doi: 10.1001/archderm.135.4.444. PMID 10206052
- [Background] Gardner ES, Reinisch L, Stricklin GP, Ellis DL. In vitro changes in non-facial human skin following CO2 laser resurfacing: a comparison study. Lasers Surg Med. 1996;19(4):379-87. doi: 10.1002/(SICI)1096-9101(1996)19:43.0.CO;2-P. PMID 8982996
- [Background] Doshi SN, Alster TS. Combination radiofrequency and diode laser for treatment of facial rhytides and skin laxity. J Cosmet Laser Ther. 2005 Mar;7(1):11-5. doi: 10.1080/14764170410003075. PMID 16020210
- [Background] Fatemi A, Weiss MA, Weiss RA. Short-term histologic effects of nonablative resurfacing: results with a dynamically cooled millisecond-domain 1320 nm Nd:YAG laser. Dermatol Surg. 2002 Feb;28(2):172-6. doi: 10.1046/j.1524-4725.2002.01112.x. PMID 11860431
- [Background] Mayoral FA. Skin tightening with a combined unipolar and bipolar radiofrequency device. J Drugs Dermatol. 2007 Feb;6(2):212-5. PMID 17373181
- [Background] Alster TS, Doshi SN, Hopping SB. Combination surgical lifting with ablative laser skin resurfacing of facial skin: a retrospective analysis. Dermatol Surg. 2004 Sep;30(9):1191-5. doi: 10.1111/j.1524-4725.2004.30370.x. PMID 15355357
- [Background] Zelickson BD, Kist D, Bernstein E, Brown DB, Ksenzenko S, Burns J, Kilmer S, Mehregan D, Pope K. Histological and ultrastructural evaluation of the effects of a radiofrequency-based nonablative dermal remodeling device: a pilot study. Arch Dermatol. 2004 Feb;140(2):204-9. doi: 10.1001/archderm.140.2.204. PMID 14967794
- [Background] Hsu TS, Kaminer MS. The use of nonablative radiofrequency technology to tighten the lower face and neck. Semin Cutan Med Surg. 2003 Jun;22(2):115-23. doi: 10.1053/sder.2003.50011. PMID 12877230
- [Background] Paul M, Blugerman G, Kreindel M, Mulholland RS. Three-dimensional radiofrequency tissue tightening: a proposed mechanism and applications for body contouring. Aesthetic Plast Surg. 2011 Feb;35(1):87-95. doi: 10.1007/s00266-010-9564-0. Epub 2010 Sep 11. PMID 20835826
- [Background] Hurwitz D, Smith D. Treatment of overweight patients by radiofrequency-assisted liposuction (RFAL) for aesthetic reshaping and skin tightening. Aesthetic Plast Surg. 2012 Feb;36(1):62-71. doi: 10.1007/s00266-011-9783-z. Epub 2011 Jul 13. PMID 21751063
- [Background] Irvine Duncan D. Nonexcisional tissue tightening: creating skin surface area reduction during abdominal liposuction by adding radiofrequency heating. Aesthet Surg J. 2013 Nov 1;33(8):1154-66. doi: 10.1177/1090820X13505862. PMID 24335016
- [Background] Boeni R. Safety of tumescent liposuction under local anesthesia in a series of 4,380 patients. Dermatology. 2011;222(3):278-81. doi: 10.1159/000327375. Epub 2011 May 24. PMID 21606638
- [Background] Nakab L, Hee CK, Guetta O. Improvements in Skin Quality Biological Markers in Skin Explants Using Hyaluronic Acid Filler VYC-12L. Plast Reconstr Surg Glob Open. 2020 Mar 27;8(3):e2723. doi: 10.1097/GOX.0000000000002723. eCollection 2020 Mar. PMID 32537370
- [Background] van Dongen JA, Langeveld M, van de Lande LS, Harmsen MC, Stevens HP, van der Lei B. The Effects of Facial Lipografting on Skin Quality: A Systematic Review. Plast Reconstr Surg. 2019 Nov;144(5):784e-797e. doi: 10.1097/PRS.0000000000006147. PMID 31688753
- [Background] Narins RS, Brandt F, Leyden J, Lorenc ZP, Rubin M, Smith S. A randomized, double-blind, multicenter comparison of the efficacy and tolerability of Restylane versus Zyplast for the correction of nasolabial folds. Dermatol Surg. 2003 Jun;29(6):588-95. doi: 10.1046/j.1524-4725.2003.29150.x. PMID 12786700
- [Background] Boroni M, Zonari A, Reis de Oliveira C, Alkatib K, Ochoa Cruz EA, Brace LE, Lott de Carvalho J. Highly accurate skin-specific methylome analysis algorithm as a platform to screen and validate therapeutics for healthy aging. Clin Epigenetics. 2020 Jul 13;12(1):105. doi: 10.1186/s13148-020-00899-1. PMID 32660606
- [Background] Fuchshuber P, Schwaitzberg S, Jones D, Jones SB, Feldman L, Munro M, Robinson T, Purcell-Jackson G, Mikami D, Madani A, Brunt M, Dunkin B, Gugliemi C, Groah L, Lim R, Mischna J, Voyles CR. The SAGES Fundamental Use of Surgical Energy program (FUSE): history, development, and purpose. Surg Endosc. 2018 Jun;32(6):2583-2602. doi: 10.1007/s00464-017-5933-y. Epub 2017 Dec 7. PMID 29218661
- See also: Ulthera White Paper. Lower Face, Submentum, and Neck — https://www.laskinmd.com/wp-content/uploads/2018/05/Ultherapy-Mechanism-of-Action-White-Paper-1002845A-1.pdf